CLINICAL TRIAL: NCT04184427
Title: Effects On Maxillary Anterior Dentition Following En- Masse Retraction Using Mini-Implants and Various Heights of Anterior Power Arm- A Randomized Controlled Trial
Brief Title: Effects on Maxillary Anterior Dentition Following En Masse Retraction Using Mini-implants and Various Heights of Anterior Power Arm.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Tahira Arif, Principal Investigator, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TArif
Record Dates: First submitted 2019-11-24; First posted 2019-12-03 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Varying Heights of Power Arm During en Masse Retraction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I (Active Comparator): 6 mm height of power arm
  Interventions: Other: Anterior Power Arm
- Group II (Experimental): 3 mm height of power arm
  Interventions: Other: Anterior Power Arm
- Group III (Experimental): 9 mm height of power arm
  Interventions: Other: Anterior Power Arm

INTERVENTIONS:
Other: Anterior Power Arm — Crimpable stainless steel hook placed on orthodontic base arch wire.
  Other Names: Anterior Retraction Hook

SUMMARY:
The controlled three dimensional movement of anterior dentition during orthodontic treatment is a desire of every orthodontist. Maxillary en masse retraction with mini implants has been reported to provide absolute anchorage thus utilizing the complete extraction spaces thereby enhancing patient's esthetics. Power arm or anterior retraction hook permits the application of force close to a desired direction thereby warranting better anterior dentition control. Various heights of power arms and proposed centre of resistance for six maxillary anterior teeth have been estimated through finite element model and also from a very limited number of clinical studies. For a set of teeth, the determination of centre of resistance is complex in actual clinical scenario and response of force applied from certain level for better anterior dentition control requires sufficient clinical evidence suggestive of further clinical studies to endow orthodontists to hasten treatment due to less time consumption during finishing stage of orthodontic treatment.

DETAILED DESCRIPTION:
This Randomized Control Trial will be conducted to compare the effects of various heights of anterior power arm on maxillary anterior dentition following en masse retraction with mini-implants by participation of thirty patients meeting eligibility criteria. The participants will be divided in three groups through software generated randomization table. Group I (control group; height of anterior power arm 6 mm), Group II and Group III (experimental groups; height of anterior power arm 3 mm and 9 mm, respectively). Ten patients will be allocated in each group. En masse retraction with mini implants and various heights of anterior power arm will be carried out immediately after bilateral maxillary first premolar extractions using continuous arch sliding mechanics. Horizontal, vertical and angular dimensions will be measured on lateral cephalograms while the transverse effects will be measured on maxillary dental cast. Both lateral cephalograms and dental casts will be obtained at two different point of time; T1, before retraction and T2, after complete extraction space closure. The data will be assessed with-in and among groups.

ELIGIBILITY:
Inclusion criteria

* Patients between ages 18-30 years.
* Good oral hygiene and healthy periodontal tissues.
* Patients having overjet ≥ 7 mm and ≤ 10 mm and overbite of 2-3 mm.
* Pt with molar relation angle's full cusp Class II requiring symmetric extractions of maxillary 1st premolars and maximum anchorage.
* Patients having coincident maxillary midline with the facial midline.

Exclusion criteria

* Patients with maxillary anterior teeth have dilacerations, fusion, hyper-cementosis, shorter roots or any other tooth anomaly.
* Patients with traumatized or impacted teeth in the anterior maxilla.
* Patients with moderate to severe crowding in maxillary and mandibular arch.
* History of bone metabolic disorders or patients receiving drugs that alter bone metabolism.
* History of systemic diseases or hormonal imbalance that hinders orthodontic tooth movement.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-06-25 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Change in maxillary central incisor sagittal dimension | Upto 1 year
  IoSV (mm), IaSV (mm), IaSV/IoSV
Change in maxillary central incisor vertical dimension | Upto 1 year
  IoPP (mm), IaPP (mm)
Change in maxillary central incisor angular dimension | Upto 1 year
  I-angle (degrees)
Change in maxillary anterior transverse dimension | Upto 1 year
  Intercanine width (mm)

CONTACTS AND LOCATIONS:
Overall Officials: Tahira Arif, Principal Investigator — Dow University of Health Sciences
Locations (1):
- Department of Orthodontics , DIEKIOHS, Dow University Of Health Sciences, Ojha Campus., Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No